CLINICAL TRIAL: NCT00928499
Title: Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
Brief Title: Trial of Continuous Versus Cyclic Stimulation in Interstim Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Karen Noblett, Division Director, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-6736
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-08

CONDITIONS: Urge Incontinence
Keywords: urge/frequency; urge incontinence; Interstim; after success Interstim planning IPG placement
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interstim - continuous (Other): Continuous stimulation
  Interventions: Device: Interstim (SNS)
- Interstim - cyclic (Other): Cyclic stimulation
  Interventions: Device: Interstim (SNS)

INTERVENTIONS:
Device: Interstim (SNS) — Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
  Other Names: Sacral nerve stimulation

SUMMARY:
Sacral Nerve Stimulation (SNS) delivers non-painful, mild electrical pulses to the sacral nerves to modulate the reflexes that influence the bladder, sphincter, and pelvic floor to improve or restore normal voiding function. Sacral nerve stimulation is indicated for refractory voiding dysfunction including urinary urgency/frequency, urinary urge incontinence, and nonobstructive urinary retention. Since its introduction, SNS has undergone significant improvements in design and application so that implantation is now a minimally invasive procedure under local and intravenous (IV) sedation. However, despite the progress made in advancing this therapy to a minimally invasive procedure, there are neither data nor guidelines on ideal program settings. The purpose of this study is to evaluate the programming parameter of cyclic versus continuous stimulation on efficacy of the therapy. If the therapy is equally efficacious at both settings, the cyclic setting has the advantage of resulting in a longer battery life.

DETAILED DESCRIPTION:
The components of SNS include a quadripolar lead wire that is placed adjacent to a sacral nerve root (typically S3), and an implantable pulse generator (IPG) that the lead wire is attached to. The IPG provides the electrical impulse and has several parameters that are amenable to adjustment including rate, strength and length of stimulation. Additionally, the stimulation can be programmed to be continuous or cyclic. If the therapy is equally efficacious at both settings, the cyclic setting has the advantage of resulting in a longer battery life. This would prolong the time interval between IPG replacements which would reduce the number of times a patient is exposed to a surgical procedure and may have a substantial impact on reducing cost to the healthcare system.

Participants will be randomized into one of two groups: either cyclic stimulation or continuous stimulation after IPG placement and will continue with this setting for four weeks. Subjects will return to the office 4 weeks post-op. They will complete a 3-day consecutive voiding diary just prior to their study visit. The subject will then undergo reprogramming to change the stimulation to the alternate pattern (from cyclic to continuous or vice versa as appropriate) keeping all other parameters the same. Subjects will be asked to return to the office 4 weeks after being switched to the alternate setting. She will complete a 3-day consecutive voiding diary just prior to the visit. The subject will also be asked their preference of mode of stimulation and the reason for their choice. After this visit, the participant will be switched to the mode of stimulation that is most efficacious for her.

ELIGIBILITY:
Inclusion Criteria:

* You are eligible to participate in this study if you have the diagnosis of urge/frequency or urge incontinence and have undergone a successful Interstim trial and are planning on proceeding with IPG placement.
* All subjects must have had a minimum of a 50% improvement of one or more of the parameters being measured on the voiding diary to be considered a candidate for implant.
* Eligibility criteria also include non-pregnant women over the age of 18 who are able to provide informed consent and are willing to accept randomization.

Exclusion Criteria:

* You are not eligible to participate in this study if:

  * you are under 18 years of age;
  * pregnant or planning to become pregnant;
  * have underlying neurological disease;
  * stress incontinence;
  * unable to read English;
  * inability to complete the voiding diary; and
  * inability to complete the follow-up visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Women's Healthcare, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinic over the course of 2 years
Pre-assignment Details: No participants were excluded.
Groups:
- Continuous Stimulation First, Then Cyclic Stimulation: Continuous stimulation first, then cyclic stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
- Cyclic Stimulation First, Then Continuous Stimulation: Cyclic stimulation first, then continuous stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
Period: Overall Study
Arm/Group | Continuous Stimulation First, Then Cyclic Stimulation | Cyclic Stimulation First, Then Continuous Stimulation
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interstim - Continuous Stimulation First, Then Cyclic Stimulation: Continuous stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
- Interstim - Cyclic Stimulation First, Then Continuous Stimulation: Cyclic stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
- Total: Total of all reporting groups
Arm/Group | Interstim - Continuous Stimulation First, Then Cyclic Stimulation | Interstim - Cyclic Stimulation First, Then Continuous Stimulation | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (12.3) | 63.4 (10.8) | 64.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Micturitions in 24 Hours
Description: Collected in the 3 day voiding diary depending on their primary diagnosis
Time Frame: After 4 weeks of stimulation a 3-day consecutive voiding diary was completed
Population: Data was insufficient to be analyzed and therefore no resulting data was collected.
Groups:
- Interstim - Continuous, Then Cyclic: Continuous stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
- Interstim - Cyclic, Then Continuous: Cyclic stimulation
  Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
Arm/Group | Interstim - Continuous, Then Cyclic | Interstim - Cyclic, Then Continuous
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Urge Incontinence Episodes in 24 Hours
Description: Collected in the 3 day voiding diary depending on their primary diagnosis
Time Frame: After 4 weeks of stimulation a 3-day consecutive voiding diary was completed
Population: Data was insufficient to be analyzed and therefore no resulting data was collected.
Arm/Group | Interstim - Continuous, Then Cyclic | Interstim - Cyclic, Then Continuous
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Interstim - Continuous, Then Cyclic: Continuous stimulation first, then cyclic stimulation Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
- Interstim - Cyclic, Then Continuous: Cyclic stimulation first, then continuous stimulation Interstim (SNS) : Randomized Controlled Trial of Continuous vs. Cyclic Stimulation in Interstim Therapy
Arm/Group | Interstim - Continuous, Then Cyclic | Interstim - Cyclic, Then Continuous
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 0/18 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No